CLINICAL TRIAL: NCT05250427
Title: Awareness, Care & Treatment In Obesity Management - An Observation in Asia Pacific
Acronym: ACTION-APAC
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-006; U1111-1266-5484 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People / Person Living with Obesity (PLwO): From online, general population consumer panels
  Interventions: Other: No treatment given
- Health Care Professionals (HCPs): HCPs treating people who have obesity
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
ACTION APAC is a cross-sectional, observational, descriptive, and exploratory survey-based study without collection of laboratory data. The study is not related to any specific treatment options or pharmaceutical product. Collection of data will be performed via quantitative online survey by a third-party vendor through existing databases/panels in APAC region.

The goal of this study is to provide insights to drive awareness around the needs of People Living with Obesity (PLwO) and Health Care Professionals (HCPs) involved in obesity treatment and management.

ELIGIBILITY:
Inclusion criteria:

People Living with Obesity

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, aged above or equal to 18 years at the time of signing informed consent
3. Lives in one of the target countries
4. Current BMI of at least 25 kg/m^2 for all countries (except Singapore which has current BMI 27 kg/m^2) based on self-reported height and weight

Health Care Professionals

1. Informed consent before any study related activities (study-related activities are any procedure related to recording/collection of data according to protocol)
2. Male or female, aged greater than or equal to 18 years at the time of signing informed consent.
3. Physician
4. Primary Care Providers (PCPs) whose specialty is Family practice, General practice, Internal Medicine
5. Non-PCP Specialties whose specialty is Endocrinologist, Cardiologist, Gastroenterologist, Obstetrics/Gynaecologist, Bariatrics/Obesity Medicine, Nutrition Specialist (physician) Orthopaedist, Aesthetics Medicine
6. Specialty is not surgeon (including bariatric or plastic surgeon)
7. Practices in the target countries
8. In clinical practice for at least 2 years
9. Spends at least 50% time in direct patient care
10. Has seen at least 100 patients in past month
11. Has seen at least 10 patients in past month who have obesity defined as: a patient with a BMI greater than or equal to 25 kg/m^2 for all countries (except Singapore which has current greater than or equal to BMI 27 kg/m^2) with or without comorbidities.

Exclusion criteria:

People Living with obesity

1. Previous participation in this study. Participation is defined as having given online consent in this study
2. Currently pregnant
3. Participates in intense fitness or body building programs
4. Has had significant, unintentional weight loss (due to major injury, illness, etc) in the past 6 months
5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Health Care Providers

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Unwillingness, inability, or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The respondent population will include people living with obesity (PLwO) and health care professionals (HCPs) involved in obesity treatment and management.
Sampling Method: Non-Probability Sample
Enrollment: 12404 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Weight loss motivators for improving health of PLwO | At the time of survey response (Day 1)
  Multi-select from defined list
Weight loss barriers for improving health of PLwO | At the time of survey response (Day 1)
  Multi-select from defined list
Weight loss management for improving health of PLwO | At the time of survey response (Day 1)
  Multi-select from defined list
Weight loss responsibility for improving health of PLwO | At the time of survey response (Day 1)
  Multi-select from defined list
Proportion of PLwO who made serious weight loss effort | At the time of survey response (Day 1)
  Number of weight loss efforts; percentage of patients
Response to weight loss discussions | At the time of survey response (Day 1)
  Single select from defined list
Attitudes towards obesity and weight management and Interactions of PLwOs with HCPs | At the time of survey response (Day 1)
  5-point Likert scales

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (9):
- Novo Nordisk Investigational Site, Dhaka, Bangladesh
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Jakarta, Indonesia
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Karachi, Pakistan
- Novo Nordisk Investigational Site, Manila, Philippines
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Novo Nordisk Investigational Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com